CLINICAL TRIAL: NCT01122043
Title: The SNEC DSAEK EndoGlide Clinical Trial
Status: Completed | Type: Observational
Sponsor: Singapore Eye Research Institute (Other)
Collaborators: UK Network Medical (Unknown)
Responsible Party: Principal Investigator, Jodhbir Mehta, Head Tissue Engineering and Stem Cell Group, Singapore Eye Research Institute
Other Study IDs: R664/14/2009; Other grant (Other Grant/Funding Number: NMRC/TCR/002 - SERI/2008 - TCR 621/41/2008])
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Bullous Keratopathy
Keywords: Endoglide; Endothelial Keratoplasty; Donor Insertion; DSAEK; Corneal Transplant; Patients with Bullous Keratopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoglide: Patients with moderate degrees of corneal decompensation from a variety of disorders which require DSAEK corneal transplantation surgery, with or without concurrent cataract surgery, to restore visual acuity.
  Interventions: Device: Endoglide

INTERVENTIONS:
Device: Endoglide — Device

SUMMARY:
The purpose of this study is to determine the clinical safety and efficacy of the EndoGlide as a donor insertion device in DSAEK surgery. The investigators hypotheses is that the Endoglide will cause less endothelial damage compared to the investigators previous technique of glide insertion but will have the same low complication rate as the previous device. Hence the investigators aim to evaluate the surgical efficacy of the EndoGlide to enable consistent double coiling of the donor lenticule in DSAEK surgery with minimal endothelial touch. Evaluate ease of insertion of the EndoGlide through a 4 to 4.5mm scleral tunnel wound. Evaluate ability of the EndoGlide to consistently effect complete wound sealing, so as to stabilize anterior chamber with an AC maintainer in position. Evaluate ease of donor pull-through from the EndoGlide chamber into the AC and to evaluate spontaneous uncoiling of the donor in the AC. Evaluate clinical efficacy and safety outcomes in EndoGlide assisted DSAEK surgery in study patients with corneal decompensation requiring DSAEK surgery, in terms of postoperative visual acuity, primary graft failure rate, donor dislocation rate, endothelial cell loss, and deturgescence of the host cornea and donor lenticule as measured by corneal thickness parameters with the Visante AS-OCT. The investigators will perfprm a prospective Phase II clinical trial using the EndoGlide for donor insertion in 100 corneal patients referred to the SNEC Corneal Clinics of the study investigators with moderate degrees of corneal decompensation from a variety of disorders which require DSAEK corneal transplantation surgery, with or without concurrent cataract surgery, to restore visual acuity.

ELIGIBILITY:
Inclusion Criteria:

1. patients presenting with corneal decompensation or bullous keratopathy requiring corneal transplantation for visual restoration and pain relief
2. Clinical diagnoses including post-surgical forms of corneal decompensation (all forms of pseudophakic and aphakic bullous keratopathy including TASS and irreversible Descemets detachment), post-laser corneal decompensation, Fuchs' and other forms of endothelial dystrophy, traumatic corneal decompensation, post-inflammatory corneal decompensation, etc.
3. Mild to moderate forms of corneal decompensation
4. patients who agree to study participation following full informed consent
5. patients who agree to adhere to the standard SNEC clinical DSAEK protocol in terms of pre and postoperative investigations and follow-up visits up to 12 months

Exclusion Criteria:

1. Severe forms or late stage presentation of corneal decompensation with severe corneal stromal scarring, unsuitable for DSAEK surgery as apposed to penetrating keratoplasty
2. patients with complex anterior segment complications precluding a successful DSAEK procedure
3. patients unkeen to participate in the clinical trial

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Bullous Keratopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Primary Graft Failure | One month

SECONDARY OUTCOMES:
Donor Graft Dislocation | One week
Endothelial Cell loss | One year

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tan, MD FRCS, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Derived] Khor WB, Mehta JS, Tan DT. Descemet stripping automated endothelial keratoplasty with a graft insertion device: surgical technique and early clinical results. Am J Ophthalmol. 2011 Feb;151(2):223-32.e2. doi: 10.1016/j.ajo.2010.08.027. Epub 2010 Dec 18. PMID 21168813